CLINICAL TRIAL: NCT02681146
Title: A Stepped-wedge Cluster Randomized Controlled Trial for Evaluating an Intervention in Patients With Stroke Tailored Education in Addition to Physiotherapist Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funded
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Phd, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMA
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: education; physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group1 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group2 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group3 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group4 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group5 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group6 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group7 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention
- Group8 (Experimental): Educational advice + physiotherapist treatment
  Interventions: Other: Multimodal intervention

INTERVENTIONS:
Other: Multimodal intervention — Educational advice + physiotherapist treatment

SUMMARY:
A stepped-wedge cluster design will be used, with the duration of the trial being 50 weeks. The 'stepped-wedge ' cluster randomised trial is a form of cross-over design with unidirectional cross-over ( from control to experimental ) but with randomisation of when each cluster undertakes this transition. In the stepped-wedge design, there is a staggered roll-out of the intervention, where the time and hence the sequence of units (clusters) that will start the intervention at each period is determined by random allocation.

The randomisation occurs before the start of the trial. All clusters start the trial in a control phase with no intervention being delivered at any site, then sequentially cross over from the control group to the intervention group, until all sites are receiving the intervention. Outcomes are measured on the study participants in all clusters at every time period, hence measurement of outcomes takes place at each step in the wedge; each cluster provides data points in the control and intervention conditions allowing each site to act as its own control.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects were all patients who had been hospitalised in 8 regional hospitals of Andalusian Health Service with acute cerebral stroke, clinically stable, presented an ischaemic or haemorrhagic aetiology and clinical symptoms of hemiplegia, were selectioned to receiving physiotherapy in hospitalisation, were assisted by a caregiver, had an adequate understanding of Spanish, and had given their written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Neurological Scale (CNS): | 8 weeks
  Measures neurological status of stroke (psychometric properties: Spearman correlation coefficient of 0.924 (95% CI: 0.896-0.951) and internal consistency by Cronbach's alpha of 0.792, N=155

SECONDARY OUTCOMES:
Trunk Control Test (TCT): | 8 weeks
  scores trunk control (psychometric properties: inter-rater reliability by Spearman's correlation coefficient r=0.76; internal consistency by Cronbach's alpha 0.83-0.86).
Motricity index (MI) of the lower and upper limbs | 8 weeks
  measures upper and lower limb strength (Spearman's correlation coefficient of 0.87 (p<0.001) for MI-LL, and of 0.88 (p<0.001) for MI-UL).
Barthel Index (BI) | 8 weeks
  scores the patient's ability to perform activities of daily living (ADL) (inter-observer reliability by Kappa indices 0.47-1.00; intra-observer reliability by Kappa indices 0.84-0.972; internal consistency by Cronbach's alpha 0.86-0.92).
Stroke Impact Scale-16 (SIS-16): | 8 weeks
  measures the deficits and physical limitations provoked by stroke (ADL, mobility and hand function) (internal consistency by Cronbach's alpha 0.87-0.95).
Modified Rankin Scale (MRS) | 8 weeks
  to score the incapacity of the patient (inter-observer reliability by Kappa indices (k=0.56 to k=0.78). Good test-re-test reliability (k=0.81 to k=0.95).
Multidimensional Scale of Perceived Social Support (MSPSS) | 8 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082